CLINICAL TRIAL: NCT05142306
Title: A Phase 1, Open-Label, Randomized Study to Evaluate Safety and Pharmacokinetics of Anti-SARS-CoV-2 Immunoglobulin (Human) Investigational Product (COVID-HIG) Administered Through Intramuscular, Subcutaneous or Intravenous Routes as a Single Dose Regimen to SARS-CoV-2 Uninfected Adults
Brief Title: A COVID-19 Study to Evaluate Safety and PK of COVID-HIG Administered Through IM, SC, or IV Routes to SARS-CoV-2 Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBS-CVH-006
Record Dates: First submitted 2021-11-30; First posted 2021-12-02 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; Coronavirus disease 2019; Severe acute respiratory syndrome coronavirus 2; immunoglobulins; intravenous; subcutaneous; intramuscular
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants in two cohorts will be enrolled and assigned equally to one of three study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- COVID-HIG Intramuscular (Experimental): Eligible subjects will be randomized to receive an 8.5mL dose of COVID-HIG by IM injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  Interventions: Biological: COVID-HIG
- COVID-HIG Subcutaneous (Experimental): Eligible subjects will be randomized to receive an 8.5mL dose of COVID-HIG by SC injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  Interventions: Biological: COVID-HIG
- COVID-HIG Intravenous (Experimental): Eligible subjects will be randomized to receive an 8.5mL dose of COVID-HIG by IV infusion.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  Interventions: Biological: COVID-HIG

INTERVENTIONS:
Biological: COVID-HIG — Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
  Other Names: NP-028

SUMMARY:
The primary objectives of this open-label trial were to evaluate the safety and pharmacokinetics (PK) of Anti-SARS-CoV-2 Immunoglobulin (Human) Investigational Product (COVID-HIG) administered intramuscularly (IM), subcutaneously (SC), or intravenously (IV) as a single dose in healthy adults 18-59 years of age with body mass index ≤35 kg/m^2. Prior studies examined IV administration, and the secondary objective of the present study was to compare PK among the three administration routes. No placebo group was included in the phase 1 randomized design. The exploratory objective was to evaluate disease severity in participants that became positive for SARS-CoV-2.

DETAILED DESCRIPTION:
Eligible participants were randomized in two cohorts to receive COVID-HIG by IM, SC or IV in a 1:1:1 ratio and were stratified based on baseline SARS-CoV-2 IgG antibody status (low seropositive/seronegative; high seropositives were excluded). Up to 36 participants were planned to be enrolled and dosed in the study. A protocol amendment truncated the study to 23 randomized participants due to the impact of high circulating SARS-CoV-2 omicron cases on enrollment and participant retention. Participants were planned to be followed through Day 85 (approximately three half-lives), but the protocol was amended to shorten the study length to Day 57 due to timeline and PK considerations. The third substantial protocol amendment change was to remove the planned pseudovirus neutralization assay from the study due to its low sensitivity, limiting the PK analysis to the S-protein binding IgG immunoassay. PK time points included predose and postdose (from end of infusion/injection) 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, Days 2, 3, 4, 6, 8, 15, 29, 43 and 57.

Nasopharyngeal swabs for SARS-CoV-2 were collected throughout the study. Per protocol, participants who became SARS-CoV-2 positive could not be assessed for PK at time points after testing positive, as the assay could not distinguish COVID-HIG from native antibodies. Participants who became SARS-CoV-2 positive during the study had disease severity assessed using an Ordinal Outcome Scale and followed via telemedicine through the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent (voluntarily signed by the participant) prior to performing study procedures.
2. Females and males 18-59 years of age.
3. Have a body mass index (BMI) less than or equal to 35.0 kg/m^2
4. Healthy, based on medical history (no chronic disease, no chronic therapy, no ongoing acute condition within four weeks prior to dosing), normal physical examination (no clinically significant findings in the opinion of the investigator), and screening laboratory assessments (no clinically significant findings in the opinion of the investigator).
5. No clinical symptoms suspicious for COVID-19 infection, as well as SARS-CoV-2 Immunoglobulin M (IgM) antibody negative and no laboratory evidence of current SARS-CoV-2 infection (i.e., reverse transcription polymerase chain reaction (RT-PCR) negative for SARS-CoV-2) at Screening.
6. Females must not be pregnant, or trying to become pregnant as demonstrated by either of the following A or B:

   A. Not of childbearing potential: surgically sterile (at least six weeks post bilateral salpingectomy, bilateral oophorectomy, or hysterectomy); or post-menopausal (history of ≥12 consecutive months without menses prior to randomization in the absence of other pathologic or physiologic causes and confirmed by follicle stimulating hormone [FSH] level ≥40 mIU/mL) OR

   B. Women of childbearing potential who are not planning to be pregnant during the study period who meet all of criteria i-iii:

   i. Negative serum pregnancy test at the Screening Visit. ii. Negative urine pregnancy test on Day 1 (a positive test will result in discontinuation from intervention).

   iii. Using one of the following highly effective methods of contraception during the study:
   1. Combined estrogen and progestogen, or progestogen-only hormonal contraception associated with inhibition of ovulation (e.g., implants, pills, patches) initiated ≥30 days prior to Study Day 1.
   2. Intrauterine device (IUD) or hormone releasing intrauterine system (IUS) inserted ≥30 days prior to Study Day 1.
7. Participant understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. Use of any investigational product within 30 days or SARS-CoV-2 monoclonal antibodies and COVID-19 convalescent plasma within 90 days prior to Screening or anticipated receipt during the study follow-up period, or participant plans to participate in another clinic study during the study period.
2. Receipt of 1 or 2 doses COVID-19 vaccine within 60 days prior to screening or during the study follow-up period.
3. SARS-CoV-2 IgG antibody levels >80 AU/mL as determined by the Diasorin LIAISON SARS-CoV-2 S1/S2 IgG antibody assay.
4. Screening clinical laboratory test result greater than the laboratory's upper limit of normal (ULN) for alanine aminotransferase (ALT), aspartate aminotransferase (AST), random glucose, total and/or direct bilirubin, blood urea nitrogen (BUN), or creatinine. Other serum chemistry parameters that are not within the reference range will not be considered exclusionary unless deemed clinically significant by the principal investigator.
5. Positive laboratory evidence of current infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV). Note: Positive anti-HCV antibody result along with a negative HCV PCR would NOT be exclusionary.
6. History of allergy or hypersensitivity to blood or plasma products or to COVID-HIG excipients (proline, PS80).
7. History of allergy to latex or rubber.
8. History of hemolytic anemia.
9. History of Immunoglobulin A (IgA) deficiency.
10. Receipt of any blood product within the past 12 months.
11. Plasma donation within 7 days or blood loss/donation (>450 mL) within 56 days of dosing.
12. History of known congenital or acquired immunodeficiency or receipt of immunosuppressive therapy (e.g., prednisone or equivalent for more than two consecutive weeks within the past three months).
13. History of thrombosis or hypercoagulable state with increased risk of thrombosis.
14. Receipt of a live vaccine within 30 days prior to screening or anticipated receipt of a live vaccine during the study period.
15. Currently pregnant, breastfeeding, or planning to become pregnant during the study.
16. History of, or suspected substance abuse problem (including alcohol).
17. Any planned elective surgery or procedure during the follow-up period that impacts study compliance.
18. Other condition which may place participant at increased risk due to participation in the study or may impact study compliance as determined by the investigator.
19. An opinion of the investigator (or designee) that it would not be in the best interest of the individual to participate in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Akintunde, MD, Study Director — Emergent BioSolutions
Locations (2):
- United States (2):
  - Qps-Mra, Llc, Miami, Florida
  - Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- COVID-HIG Intramuscular (IM): Eligible subjects will be randomized to receive an 8.5mL dose of COVID-HIG by IM injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  COVID-HIG: Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
- COVID-HIG Subcutaneous (SC): Eligible subjects will be randomized to receive an 8.5mL dose of COVID-HIG by SC injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  COVID-HIG: Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
- COVID-HIG Intravenous (IV): Eligible subjects will be randomized to receive an 8.5mL dose of COVID-HIG by IV infusion.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  COVID-HIG: Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
Period: Overall Study
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Started | 7 | 8 | 8
Safety Population | 7 | 8 | 7
Completed | 7 | 8 | 7
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data is from the safety population which includes all subjects who received any amount of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV) | Total
Number analyzed (Participants) | 7 | 8 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (9.7) | 36.3 (13.0) | 32.4 (9.2) | 38.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 2 | 10
  Male | 5 | 2 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 3 | 12
  Not Hispanic or Latino | 3 | 3 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 8 | 7 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 172.57 (3.88) | 163.31 (7.94) | 170.14 (6.28) | 168.43 (7.30)
Baseline weight [Mean (Standard Deviation); unit: kilograms] | 86.51 (12.95) | 67.29 (13.78) | 73.69 (7.62) | 75.44 (13.96)
Baseline body mass index [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 28.94 (3.48) | 25.09 (4.12) | 25.56 (3.49) | 26.46 (3.96)
Baseline SARS-CoV-2 Antibody Status [Count of Participants; unit: Participants] — As measured using the Diasorin LIAISON S1/S2 IgG assay. Seronegative indicates no detectable antibody (<15 AU/mL; <LLOQ). Seropositive indicates detectable antibody ≥15, but ≤80 AU/mL. Subjects with antibody level >80 AU/mL were excluded from the study (as per exclusion criteria #3).
  Participants
    Seronegative | 4 | 4 | 4 | 12
    Seropositive | 3 | 4 | 3 | 10
Enrollment per Study Site [Count of Participants; unit: Participants]
  US6001 (Miami, FL) | 4 | 5 | 3 | 12
  US6002 (Springfield, MO) | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events (AEs) up to 72 Hours Post-dosing
Description: Number of participants with AEs and severity of AEs up to 72 hours post-dosing.
Time Frame: 72 hours
Population: Safety population includes all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- COVID-HIG Intramuscular (IM): Eligible participants will be randomized to receive an 8.5mL dose of COVID-HIG by IM injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  COVID-HIG: Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
- COVID-HIG Subcutaneous (SC): Eligible participants will be randomized to receive an 8.5mL dose of COVID-HIG by SC injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  COVID-HIG: Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
- COVID-HIG Intravenous (IV): Eligible participants will be randomized to receive an 8.5mL dose of COVID-HIG by IV infusion.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
  COVID-HIG: Anti-SARS-CoV-2 Immunoglobulin (Human) [COVID-HIG] is a purified liquid immunoglobulin G (IgG) preparation
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
Participants | 2 | 1 | 2

2. Primary Outcome: Participants With Adverse Events That Led to Discontinuation or Temporary Suspension of Study Treatment
Description: Number of participants and severity of AEs that led to discontinuation or temporary suspension of study treatment.
Time Frame: Day 1
Population: Safety population includes all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
Participants | 0 | 0 | 0

3. Primary Outcome: Participants With AEs and SAEs After Study Treatment
Description: Number of participants with adverse events (AEs) and serious adverse events (SAEs) up to 56 days post-administration of a single dose of COVID-HIG.
Time Frame: Day 0 to Day 57
Population: Safety population includes all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
Participants
  Number of participants with any AE | 6 | 3 | 4
  Number of participants with any SAE | 0 | 0 | 0

4. Primary Outcome: Total Number of AEs and SAEs After Study Treatment
Description: Number of adverse events (AEs) and serious adverse events (SAEs) in all participants reporting AEs/SAEs up to 56 days post-dosing.
Time Frame: Day 0 to Day 57
Population: Safety population includes all participants who received any amount of study treatment.
Measure: Number; unit: Events
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
Events
  Total number of adverse events (AEs) for all participants reporting AEs | 9 | 5 | 9
  Total number of SAEs for all participants reporting SAEs | 0 | 0 | 0

5. Primary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to the Last Quantifiable Concentration (AUC0-last) of SARS-CoV-2 Antibodies After Dose of COVID-HIG
Description: The area under the concentration-time curve from time 0 to the last quantifiable concentration of SARS-CoV-2 binding IgG antibodies after COVID-HIG dose. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: The PK population included all subjects who received COVID-HIG and had an adequate set of evaluable PK samples (a suitable predose sample and at least one measurable postdose sample, with samples occurring after a positive SARS-CoV-2 test result excluded).
Measure: Geometric Mean (95% Confidence Interval); unit: h*Alliance Units (AU)/mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
h*Alliance Units (AU)/mL | 6435.44 [1889.47 to 21918.78] | 9560.60 [3382.99 to 27018.99] | 11883.46 [6891.36 to 20491.83]

6. Primary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time (AUC) From Time 0 to Infinity (AUC0-inf) After Dose of COVID-HIGIV
Description: Area under the concentration-time curve from time 0 to the last quantifiable concentration plus the additional area extrapolated to infinity of SARS-CoV-2 binding IgG antibodies after COVID-HIG dose. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 2 | 3 | 4
h*AU/mL | 8042.38 [2561.73 to 25248.55] | 6875.52 [5521.48 to 8561.60] | 19212.18 [7569.07 to 48765.28]

7. Primary Outcome: Pharmacokinetics Parameter of Maximum Observed Concentration (Cmax) of SARS-CoV-2 Antibodies Observed After Dose of COVID-HIG
Description: The Cmax of SARS-CoV-2 binding IgG antibodies observed after COVID-HIG dose. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
AU/mL | 17.02 [8.00 to 36.24] | 16.24 [7.62 to 34.65] | 56.88 [30.41 to 106.39]

8. Primary Outcome: Pharmacokinetics Parameter of Time at Which Cmax Occurs After Dose of COVID-HIG
Description: Time at which Cmax occurs (Tmax) after COVID-HIG dose. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 7 | 8 | 7
hours | 174.71 (221.13) | 201.01 (213.76) | 1.53 (0.53)

9. Primary Outcome: Pharmacokinetics Parameter of Trough Concentration of SARS-CoV-2 Antibodies Observed 28 Days After Dose (Cmin28d) of COVID-HIG
Description: The observed trough concentration of SARS-CoV-2 binding IgG antibodies 28 days after COVID-HIG dose. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, and Day 29.
Time Frame: Day 1 to Day 29
Population: The PK population included all subjects who received COVID-HIG and had an adequate set of evaluable PK samples up to Day 29.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 4 | 6 | 5
AU/mL | 3.67 [0.00 to 15928.95] | 7.55 [2.36 to 24.19] | 8.15 [5.58 to 11.91]

10. Secondary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to 28 Days (AUC0-28d) After Dose of COVID-HIG.
Description: AUC from time 0 to 28 days of SARS-CoV-2 binding IgG antibodies after COVID-HIG dose. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, and Day 29.
Time Frame: Day 1 to Day 29
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 4 | 6 | 5
h*AU/mL | 14610.82 [3072.14 to 69487.73] | 14624.92 [4470.66 to 47842.64] | 12182.14 [6935.59 to 21397.55]

11. Secondary Outcome: Pharmacokinetics Parameter of Area Under the Concentration-time Curve (AUC) From Time 0 to 14 Days After Dose of COVID-HIG
Description: AUC from time 0 to 14 days (AUC0-14d) of SARS-CoV-2 binding IgG antibodies after COVID-HIG. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, and Day 15.
Time Frame: Day 1 to Day 15
Population: The PK population included all subjects who received COVID-HIGIV and had an adequate set of evaluable PK samples up until Day 15.
Measure: Geometric Mean (95% Confidence Interval); unit: h*AU/mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 5 | 7 | 7
h*AU/mL | 12057.04 [3700.79 to 39281.36] | 11118.31 [3465.31 to 35672.65] | 11883.46 [6891.36 to 20491.83]

12. Secondary Outcome: Pharmacokinetics Parameter of Apparent Terminal Elimination Half-life (T1/2) After Dose of COVID-HIG
Description: The apparent terminal elimination half-life (T1/2) after dose of COVID-HIG. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: The PK population included all subjects who received COVID-HIG and had an adequate set of evaluable PK samples.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 2 | 3 | 4
hours | 505.50 (128.13) | 535.70 (61.09) | 673.90 (356.02)

13. Secondary Outcome: Pharmacokinetics Parameter of Systemic Clearance (CL) After Dose of COVID-HIG
Description: The systemic clearance (CL) of SARS-CoV-2 binding IgG antibodies after dose of COVID-HIG. . Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: The PK population included all subjects who received COVID-HIG and had an adequate set of evaluable PK samples.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 2 | 3 | 4
mL/h | 0.0010 (0.0000) | 0.0010 (0.0000) | 0.0010 (0.0006)

14. Secondary Outcome: Pharmacokinetic Parameter of Volume of Distribution (Vz) After Dose of COVID-HIG
Description: The volume of distribution (Vz) of SARS-CoV-2 binding IgG antibodies after dose of COVID-HIG. Data for PK calculations was collected: pre-dose, and post-dose at: 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, Day 3, Day 4, Day 6, Day 8, Day 15, Day 29, Day 43, and Day 57.
Time Frame: Day 1 to Day 57
Population: The PK population included all subjects who received COVID-HIG and had an adequate set of evaluable PK samples.
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
Number analyzed (Participants) | 2 | 3 | 4
mL | 0.75 [0.32 to 1.75] | 0.93 [0.67 to 1.28] | 0.35 [0.27 to 0.45]

15. Other Pre Specified Outcome: Comparative Bioavailability: Area Under the Concentration-time Curve (AUC) From Time 0 to Last (AUC0-last) Ratios Between Administration Routes
Description: AUC0-last ratios (bioavailability) compared between routes for comparable dose levels (COVID-HIG IM to SC; SC to IV; and IM to IV). Least square mean estimates and 90% confidence intervals were derived from ANOVA model with AUC0-last as dependent variable and administration route as fixed effect. Comparative bioavailability was defined as within [80%, 125%].
Time Frame: Day 1 to Day 57
Population: The PK population included all subjects who received COVID-HIG and had an adequate set of evaluable PK samples. In each arm, there were n=7 in the COVID-HIG IM arm, n=8 in the COVID-HIG SC arm and n=7 in the COVID-HIG IV arm. The overall participants analyzed per group as indicated in this bioavailability comparison is the sum of each of the respective groups indicated in the title/description.
Measure: Number (90% Confidence Interval); unit: ratio
Groups:
- COVID-HIG IM Versus SC: Comparison between eligible subjects randomized to receive an 8.5mL dose of COVID-HIG by intramuscular (IM) or subcutaneous (SC) injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
- COVID-HIG IM Versus IV: Comparison between eligible subjects randomized to receive an 8.5mL dose of COVID-HIG by intramuscular (IM) or intravenous (IV) injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
- COVID-HIG SC Versus IV: Comparison between eligible subjects randomized to receive an 8.5mL dose of COVID-HIG by subcutaneous (SC) or intravenous (IV) injections.
  COVID-HIG: COVID-HIG is a purified immunoglobulin G (IgG) liquid preparation containing antibodies (including neutralizing antibodies) to SARS-CoV-2.
Arm/Group | COVID-HIG IM Versus SC | COVID-HIG IM Versus IV | COVID-HIG SC Versus IV
Number analyzed (Participants) | 15 | 14 | 15
ratio | 0.67 [0.25 to 1.82] | 0.54 [0.19 to 1.51] | 0.80 [0.30 to 2.17]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 (Dosing Day) through Day 57 or early withdrawal.
Description: Adverse events were unsolicited.
Arm/Group | COVID-HIG Intramuscular (IM) | COVID-HIG Subcutaneous (SC) | COVID-HIG Intravenous (IV)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 3/8 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVID-HIG Intramuscular (IM) (N=7) | COVID-HIG Subcutaneous (SC) (N=8) | COVID-HIG Intravenous (IV) (N=7)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Bacterial Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT05142306/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT05142306/SAP_001.pdf
  • Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT05142306/ICF_002.pdf